CLINICAL TRIAL: NCT03679598
Title: A First in Class Disease Modifying Therapy to Treat Alpha-1 Antitrypsin Deficiency a Genetically Linked Orphan Disease
Brief Title: Alvelestat (MPH966) for the Treatment of ALpha-1 ANTitrypsin Deficiency
Acronym: ATALANTa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Mereo BioPharma (Industry); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Mark Dransfield, MD, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-300002338; 4UH3TR002450-02 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2018-09-20 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Alpha-1 Antitrypsin Deficiency (AATD); Pi*ZZ, Pi*SZ, Pi*Null, Another Rare Phenotype/Genotype Known to be Associated With Either Low or Functionally Impaired AAT Including F or I Mutations; Emphysema or COPD
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: randomized (1:1), placebo-controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alvelestat (MPH966) (Active Comparator): Alvelestat (MPH966) 120mg (4 30mg tablets) twice daily by mouth for 12 weeks
  Interventions: Drug: Alvelestat (MPH966)
- Placebo (Placebo Comparator): 4 Placebo tablets twice daily by mouth for 12 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alvelestat (MPH966) — Alvelestat was developed as treatment for lung diseases like Chronic Obstructive Pulmonary Disease. Alevelestat works by blocking certain proteins in the body that are responsible for inflammation and damage to the lungs that can lead to COPD symptoms.
  Arms: Alvelestat (MPH966)
Other: Placebo — Placebo is a pill or tablet that does not contain any study drug.
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, double-blind, randomized (1:1), placebo-controlled, 12-week, proof-of-concept study to evaluate the safety and tolerability as well as the mechanistic effect of oral administration of alvelestat (MPH966) in subjects with confirmed AATD defined as Pi*ZZ, Pi*SZ, Pi*null, or another rare phenotype/genotype known to be associated with either low (serum AAT level <11 μM or <57.2 mg/dL) or functionally impaired AAT including "F" or "I" mutations.

DETAILED DESCRIPTION:
Alpha-1 antitrypsin deficiency (AATD) is the most common genetic cause of chronic obstructive pulmonary disease (COPD) and early-onset emphysema. AATD is characterized by low AAT levels; leading to excessive neutrophil elastase (NE) mediated lung destruction. Current treatment requires the periodic infusion of pooled AAT derived from human plasma, but this therapeutic approach (termed augmentation) does not definitively slow the rate of emphysema progressionlung function decline and is very expensive. In addition, it is not clear that the currently recommended dose for augmentation fully controls lung inflammation and destruction. Alvelestat (MPH966, formerly AZD9668) is a potent, selective, and reversible, oral inhibitor of human NE. Suppression of NE is expected to reduce lung damage and may slow disease progression. This study is to establish proof of clinical concept by investigating the mechanistic effect and safety of alvelestat (MPH966) in patients with AATD.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if ALL of the following criteria apply:

1. Capable of giving signed informed consent as described in Appendix 3, which includes compliance with the requirements and restrictions listed in the informed consent form and in this protocol
2. Age ≥18 and ≤80 years
3. Patients with a confirmed diagnosis of AATD: Pi*ZZ, Pi*SZ, Pi*null, or another rare phenotype/genotype known to be associated with either low (serum AAT level <11 μM or <57.2 mg/dL) or functionally impaired AAT including "F" or "I" mutations.
4. FEV1 ≥25% predicted
5. Patients will be eligible if they are either a) are not currently receiving augmentation treatment and have not received augmentation in the 12 weeks prior to screening or b) have received weekly infusions of augmentation at 60 mg/kg for at least 12 weeks prior to screening and intend to continue augmentation through the study period.
6. Male or female sex a. Male participants must agree to use a highly effective contraception as detailed in Appendix 5 during the treatment period and for at least 4 days after the last dose of study treatment and refrain from donating sperm during this period b. Female participants are eligible to participate if not pregnant; not breastfeeding; and at least one of the following conditions is met: i. Not a woman of childbearing potential as defined in Appendix 5 OR ii. A woman of childbearing potential who agrees to follow the contraceptive guidance in Appendix 5. During the treatment phase and for at least 4 days after the last dose of study medication.

Exclusion Criteria:

Participants are excluded from the study if ANY of the following criteria apply:

Excluded Medical Conditions

1. Subjects with Pi*MZ, Pi*FM, Pi*MS, Pi*SS, or other AATD phenotypes/genotypes not known to be independently associated with emphysema.
2. Any clinically diagnosed lung disease other than COPD such as diffuse interstitial lung diseases, cystic fibrosis, or clinically significant bronchiectasis as determined by the Investigator
3. Acute exacerbation of underlying lung disease requiring oral steroids and/or antibiotics within 4 weeks of baseline
4. Acute or chronic hepatitis, including hepatitis B, hepatitis C (positive serologies, including hepatitis B and C antibody)
5. HIV infection or other immunodeficiency or with an absolute neutrophil count ≤1.0 × 109/L
6. Abnormal liver biochemistry (alanine aminotransferase, aspartate aminotransferase, gamma-glutamyl transferase) >1.5 × upper limit of normal or total bilirubin > upper limit of normal (unless Gilbert's disease with normal conjugated bilirubin)
7. Any of the following laboratory abnormalities are present at baseline:

   1. Platelet count <150×109/L
   2. Serum albumin ≤ 3.5 g/dL
   3. INR ≥1.2
   4. CPK ≥ ULN.
8. History or current evidence of cirrhosis (on biopsy or imaging), esophageal varices, ascites or hepatic encephalopathy.
9. Evidence of other forms of chronic liver disease based on diagnostic testing as per the guidelines (i.e. autoimmune liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson's disease, Hemochromatosis or iron overload).
10. Patients with nonalcoholic fatty liver disease (NAFLD) as diagnosed by any imaging modality (or use of drugs associated with NAFLD for more than 2 weeks in the year prior to screening).
11. Subjects with a history of significant alcohol consumption for a period of more than 3 consecutive months within 1 year prior to screening, defined as average of >20g/ day in female subjects and >30g/ day in male subjects.
12. Fibrosis-4 (FIB-4) score >3.25
13. Any of the following cardiovascular conditions within 6 months prior to the screening visit:

    1. Myocardial infarction or unstable angina
    2. Coronary artery bypass surgery, balloon angioplasty, percutaneous coronary intervention, or carotid revascularization procedure
    3. Uncontrolled hypertension
    4. Stroke or transient ischemic attack
14. Congestive heart failure (New York Heart Association III/IV) with left ventricular ejection fraction < 40%
15. Any clinically significant 12-lead electrocardiogram abnormalities at screening or baseline, including corrected QT interval by Fridericia's correction method >450 ms or history of significant cardiac dysrhythmia, including long QT syndrome
16. History of cancer within the last 5 years, except for well-treated basal cell carcinoma and squamous cell carcinoma of the skin
17. Other documented comorbidities or laboratory abnormalities that in the opinion of the Investigator could affect the outcome of the study assessments, participant safety, or ability of the participant to comply with the requirements of the protocol

    Excluded Prior/Concomitant Therapy
18. Daily use of prednisone (>10mg daily), or other systemic glucocorticoids at comparable or higher equivalent dose, or use of other immunosuppressant therapies are prohibited
19. Immunomodulating monoclonal antibodies within 6 months prior to screening are prohibited
20. Daily use of non-steroidal anti-inflammatory drugs (NSAIDs) is prohibited. Daily use of acetaminophen up to 2 g per day and aspirin up to 325 mg per day is permitted.
21. Initiation of drugs known for hepatotoxic potential within the 28 days prior to screening including but not limited to: statins, NSAIDS, amoxicillin/clavulanate, PDE inhibitors (theophylline, roflumilast), and anti-epileptics. Subjects on established treatment for more than 28 days prior to screening will not be excluded. Requirement for medications mainly metabolized by CYP2C9 and with narrow therapeutic index (eg, warfarin, phenytoin) is prohibited

    Excluded Prior/Concurrent Clinical Study Experience
22. Participation in any clinical investigation using medical devices or non-biologic treatments within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to the initial dosing (or longer if required by local regulations) is prohibited
23. Participation in any clinical investigation using biologic treatment within 6 months of screening is prohibited
24. Previous participation in a gene therapy study for AATD at any time is prohibited

    Other Exclusions
25. History of hypersensitivity to alvelestat (MPH966) or any of its excipients or the class of neutrophil elastase inhibitors
26. Known hypersensitivity to medications used in the study procedures (e.g. midazolam, fentanyl, and lidocaine for bronchoscopy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark T Dransfield, MD, Principal Investigator — University of Alabama at Birmingham
Locations (10):
- United States (10):
  - The University of Alabama at Birmingham Lung Health Center, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Columbia University, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alvelestat (MPH966) | Placebo
Started | 32 | 31
Completed | 30 | 31
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvelestat (MPH966) | Placebo | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (14.0) | 54.6 (11.9) | 53.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 30 | 30 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 31 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Alpha-1 antitrypsin Genotype [Count of Participants; unit: Participants]
  Pi*NN | 2 | 3 | 5
  Pi*SZ | 6 | 4 | 10
  Pi*ZZ | 22 | 24 | 46

OUTCOME MEASURES:

1. Primary Outcome: Within-individual % Change in Plasma Desmosine/Isodesmosine
Description: To evaluate the effect of alvelestat (MPH966) administered twice daily (bid) for 12 weeks on blood markers of within-individual % change in plasma desmosine/isodesmosine will be measured.
Time Frame: baseline, week 12
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Alvelestat (MPH966) | Placebo
Number analyzed (Participants) | 29 | 30
% change | 10.0619 (27.8489) | 8.5627 (29.2973)

2. Primary Outcome: Numbers and % of Subjects Who Experience at Least 1 Treatment-emergent Adverse Event
Description: To evaluate the safety and tolerability of alvelestat (MPH966) administered twice daily (bid) for 12 weeks treatment numbers and % of subjects who experience at least 1 treatment-emergent adverse event (TEAE) will be measured.
Time Frame: baseline, week 16
Measure: Count of Participants; unit: Participants
Arm/Group | Alvelestat (MPH966) | Placebo
Number analyzed (Participants) | 32 | 31
Participants | 25 | 23

3. Secondary Outcome: Blood Pharmacodynamic Markers of Neutrophil Activation and Elastase Activity. Change From Baseline in the Following Outcomes at End of the Treatment Within Patient and Compared to Placebo
Description: To evaluate the effect of Alvelestat (MPH966) on other blood pharmacodynamic markers of neutrophil activation and elastase activity including plasma desmosine/isodesmosine (change compared to placebo; within-individual change is the primary outcome), plasma Aa-Val-360, serum NE activity, plasma proteinase 3, plasma cathepsin B, plasma CRP, plasma IL-6, plasma IL-8, plasma IL-1b, plasma RANTES, plasma LTB4, plasma MMP9, plasma MMP12, plasma MPO, and plasma PGP.
Time Frame: baseline, week 12
Measure: Mean (Standard Deviation); unit: ng/ mL
Arm/Group | Alvelestat (MPH966) | Placebo
Number analyzed (Participants) | 29 | 30
ng/ mL
  Plasma desmosine/isodesmosine | 0.0307 (0.1012) | 0.0047 (0.0817)
  Plasma Aa-Val-360 | -1.6279 (4.1028) | -0.9937 (4.3209)
  Serum NE | -16.7926 (41.1503) | 3.9660 (19.4462)
  Plasma proteinase 3 | 1.9412 (59.2846) | -10.6390 (38.6356)
  Plasma cathepsin B | 7.2882 (24.9583) | -1.1086 (14.6929)
  Plasma CRP | -0.0247 (1.1066) | -0.1975 (1.6880)
  Plasma IL-6 | 0.3417 (2.1615) | -0.3730 (2.7773)
  Plasma IL-8 | -0.2955 (2.9877) | 0.2386 (0.8844)
  Plasma IL-1b | 0.0962 (0.3819) | 0.1137 (0.5218)
  Plasma RANTES | 0.0903 (3.9356) | 0.0652 (6.4001)
  Plasma LTB4 | -369.093 (11118.482) | 170.2617 (1380.099)
  Plasma MMP9 | -2.8218 (18.6240) | 2.6188 (8.7639)
  Plasma MMP12 | -1.0733 (8.0076) | -0.0940 (1.6722)
  Plasma MPO | -4516.01 (24994.15) | 3156.253 (13798.49)
  Plasma PGP | -0.6619 (3.8013) | -0.0139 (0.5418)

ADVERSE EVENTS:
Time Frame: Baseline to week 16
Description: Adverse events of special interest include liver function abnormalities, corrected QT interval/cardiac, infections, and neutropenia. Treatment-emergent AEs (TEAEs) are defined as any AE occurring on or after the first dose of study medication. AEs will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), and summarized by system organ class and preferred term.
Arm/Group | Alvelestat (MPH966) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/31
Other Adverse Events (participants affected / at risk) | 25/32 | 23/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvelestat (MPH966) (N=32) | Placebo (N=31)
Headache (Nervous system disorders) | 12 (15) | 7 (7)
Migraine (Nervous system disorders) | 2 (2) | 2 (3)
Restless legs syndrome (Nervous system disorders) | 1 (2) | 0 (0)
Sinus headache (Nervous system disorders) | 2 (2) | 0 (0)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Vaginal infection (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 5 (5)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT03679598/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT03679598/SAP_003.pdf